Title of the study: Effect of Adipose Derived Stem Cells on Survival of Fat as Filler

Date of the document: January 1, 2019

## **Investigators and study group:**

## Osama Hussein Roshdy MD, PhD

Professor of Dermatology, Dermatology Department, Faculty of Medicine, Alexandria University, Egypt.

## Wafaa Ibrahim Abdullah MD, PhD

Professor of Dermatology, Dermatology Department, Faculty of Medicine, Alexandria University, Egypt.

### Carmen Ibrahim Farid Mohammed Amin MD, PhD

Professor of Dermatology, Dermatology Department, Faculty of Medicine, Alexandria University, Egypt.

## Radwa Ali Mehana, MD, PhD

Assistant Professor of Physiology, Physiology Department, Faculty of Medicine, Alexandria University, Egypt.

# Nader Hussein Lotfy Bayoumi. MD, PhD, FRCS (Glasgow)

Professor of Ophthalmology, Ophthalmology Department, Faculty of Medicine, Alexandria University, Egypt.

# Aliaa Ismail, MD, PhD

Assistant Lecturer of Dermatology, Dermatology Department, Faculty of Medicine, Alexandria University, Egypt.

#### INTRODUCTION

Skin aging is a complex biological process that can be categorized into either extrinsic or intrinsic aging. Intrinsic aging is an inherent degenerative process caused by decreased proliferative capacity leading to cellular senescence. Extrinsic aging is caused by factors such as UV radiations, smoking and alcohol consumption.<sup>(1,2)</sup>

The physiological changes associated with aging of the skin are manifested in xerosis, dramatic loss of skin elasticity due to damage to collagen and elastin fibers; as well as barrier function, modification of rhytides and deficiencies in the regenerative property of the skin. All of which ultimately result in thinning of the skin, malar fat atrophy and pigmentary changes.<sup>(3)</sup>

Aging skin undergoes thinning of the epidermis that is caused by reduction of vascularity and hydration. On average, the thickness of the epidermis is reduced by about 6.4% during each decade of life.<sup>(4)</sup>

Skin aging effects can be assessed based on the skin appearance (texture and roughness, fine lines and wrinkles), structure, elasticity, hydration and barrier function. Many new non-invasive or minimally invasive bioengineering advances in recent years have enabled the quantitative analysis of skin properties during the aging process.<sup>(5)</sup>

There are an increasing number of treatment modalities to improve the appearance of aging skin including dermal fillers, injectable botulinum toxin, laser, chemical peeling and a diverse of topical agents including topical retinoid. (6)

Autologous fat grafting or lipo injection containing stromal vascular fraction (SVF) acts like ideal soft tissue filler for facial filling and rejuvenation. (4) It leads to progressive improvement of the skin texture, elasticity, and color over a few

months, therefore adipose tissue seems to be not only a simple filler but also a dynamic filler with two types of different and supplementary effects, the volumetric effect and the regenerative effect.<sup>(7)</sup>

Recently, adult stem cells such as mesenchymal stem cells (MSCs) have been used in variable dermatologic conditions due to its regenerative properties such as wound healing, rejuvenation, acne scar and hair fall treatment. Different types of MSCs could be derived from different tissues as for example; bone marrow stem cells (BMSCs), adipose tissue-derived stem cells (ADSCs), and skin-derived stem cells (SDSCs).<sup>(8)</sup>

Adipose tissue derived stem cells are currently favorable compared to other types of adult stem cells as the procedure is easy, safe with minimal donor site morbidity. The process of obtaining a considerable amount of adipose tissues sufficient to use in skin regeneration is highly appealing due to its relative availability and accessibility. They secrete variable growth factors that affect surrounding environment as vascular endothelial growth factor (VEGF), platelet derived growth factor (PDGF), insulin like growth factors (IGF) and others. (9)

Cell assisted lipotransfer (CAL) is a technique that combines aspirated fat with concentrated ADSCs in the stromal vascular fraction (SVF) of the lipoaspirate. This technique could enhance the survival rate of the transplanted fat and leads to better cosmetic improvement.<sup>(8)</sup>

# AIM OF THE WORK

The aim of this work is to evaluate the effect of Adipose Derived Stem Cells on Survival of Fat as Filler

#### **PATIENTS**

The current study will be carried out on 15 healthy female participants recruited from the Outpatient Clinic of the Dermatology Department of Alexandria Main university hospital.

#### **Inclusion criteria:**

- 1. Clinically diagnosed facial skin aging.
- 2. Glogau photoaging score II and III.
- 3. Body mass index ≥20 with adequate abdominal or other subcutaneous adipose tissue accessible for lipoaspiration.

#### **Exclusion criteria:**

- 1. History of keloid formation.
- 2. Any coincidental chronic illness (e.g. metabolic, autoimmune or endocrinal) or malignancy.
- 3. Any bleeding or coagulation disorder or recent use of anticoagulant therapy.
- 4. Active infection.
- 5. History of any previous aesthetic procedure on the face within the past 6 months.
- 6. History of intake of anti-aging systemic or topical medications within the previous 3 months.

An informed consent for both participations in the study and photography will be taken from all participants prior to the onset of the study after full explanation of the procedure and its follow up steps. Patients will have to sign to committing to the study protocol, using sun protection, and abstaining from using or doing any anti-ageing steps during the study period.

#### **METHODS**

#### All participants will be subjected to:

- 1. Full history taking including personal, family, medical and drug history.
- 2. History of any previous aesthetic procedures on the face.
- 3. BMI calculation. (10)
- 4. Baseline assessment of facial skin ageing will be done using the following techniques:
  - Base line standardized digital photography of the face before the procedure and in each follow up visit.
  - Assessment of degree of improvement using Hollowness severity rating scale: 0: no visible hollowness, 1: mild Hollowness, 2: moderate H, 3: severe Hollowness on serial photography.
  - Assessment of trans-epidermal water loss (TEWL) and skin hydration using noninvasive probe (Dermal measurement system EDS12, UK) on both temple regions of the head. (13)
  - Measurement of epidermal, dermal and hypodermal thickness using UBM (Ultrasound Bio microscopy) on both temple regions of the head.<sup>(14)</sup>

# Lipoaspiration for preparation of ADSC will be done according to the following technique: $\sp(7)$

Under local anesthesia using strict aseptic technique, a small incision will be done in the lateral aspect of the thigh or lower abdomen, through which the infiltration cannula will be introduced to inject the local anesthetic solution using the wet technique. This will be followed 15 minutes later by lipo-aspiration of (50 ml fat) using a blunt tipped cannula under the negative suction pressure of a 60 ml syringe.

 Autologous adipose tissue derived stem cells (At-ADSCs) will be separated from the lipo-aspirate using enzymatic digestion and

- differential centrifugation in the Center of Excellence for Research in Regenerative Medicine and its Application (CERRMA), Alexandria Faculty of Medicine.
- Viability of collected cells will be checked using trypan blue stain. (15) Characterization of the isolated ADSCs population will be performed by flow cytometry to check for specific cell surface CD antigens (CD 90 and CD 34) in three independent cases in triplet. (7)

Aspiration of 75 ml of fat followed by preparation of At-ADSCs from 25 ml.

• One temporal region is randomly selected as control to receive the required volume of fat via subcutaneous injection using blunt cannula. The other side receive equal volume of fat enriched with ADSCs in SVF.

#### Follow up and evaluation:

- Early assessment of trans-epidermal water loss (TEWL) and skin hydration will be carried out a week after the procedure.
- All participants will be followed up six months after the procedure. Follow up will entail using the same base line assessment steps to detect the effects of treatment. Side effects reported by the participants will be recorded.
- Assessment of the participants and the photos will be carried out by a blinded investigator to the half treated and the before versus after photos.
- A visual analog scale, <sup>(16)</sup> will be used to assess participants' satisfaction by the treatment

| Research on human | or human products: |
|---|---|
| • | ve study: informed consent will be taken from patients. In etent patients the informed consent will be taken from the |
| Retrospec | ctive study: confidentiality of records will be considered. |
| and for research<br>out except with | nomic material: informed consent for DNA / genomic test will be taken from patients. No further test will be carried further approval of committee and patients. If the samples de Egypt the researcher will be responsible for transportation proval. |
| All drugs of Health. | used in the research are approved by the Egyptian Ministry |
| Research on animal: | |
| The anim | al species are appropriate for the test. |
| After test disposed. | , if animal will suffer, it will be euthanized and properly |
| After ope | eration, it will have a proper postoperative care. |

# **RESULTS**

The results obtained will be tabulated, statistically analyzed and findings will be illustrated using tables and figures.

# **DISCUSSION**

The results obtained will be discussed in view of achievement of the aim of the work and compared with other findings in literature.

#### REFERENCES

- 1. Makrantonaki E, Zouboulis CC. Molecular mechanisms of skin aging: state of the art. Ann N Y Acad Sci 2007; 1119:40-50.
- 2. Yaar M, Gilchrest BA. Photoageing: mechanism, prevention and therapy. Br J Dermatol 2007; 157(5):874-87.
- 3. Zouboulis CC, Makrantonaki E. Clinical aspects and molecular diagnostics of skin aging. Clin Dermatol 2011; 29(1):3-14.
- 4. Gaur M, Dobke M, Lunyak VV. Mesenchymal Stem Cells from Adipose Tissue in Clinical Applications for Dermatological Indications and Skin Aging. Int J Mol Sci 2017; 18(1):13-7.
- 5. Hahn HJ, Jung HJ, Schrammek-Drusios MC, Lee SN, Kim JH, Kwon SB, et al. Instrumental evaluation of anti-aging effects of cosmetic formulations containing palmitoyl peptides, Silybum marianum seed oil, vitamin E and other functional ingredients on aged human skin. Exp Ther Med 2016; 12(2):1171-6.
- 6. Tierney EP, Hanke CW. Recent advances in combination treatments for photoaging: review of the literature. Dermatol Surg 2010; 36(6):829-40.
- 7. Rigotti G, Charles-de-Sa L, Gontijo-de-Amorim NF, Takiya CM, Amable PR, Borojevic R, et al. Expanded Stem Cells, Stromal-Vascular Fraction, and Platelet-Rich Plasma Enriched Fat: Comparing Results of Different Facial Rejuvenation Approaches in a Clinical Trial. Aesthet Surg J 2016; 36(3):261-70.
- 8. Salibian AA, Widgerow AD, Abrouk M, Evans GR. Stem cells in plastic surgery: a review of current clinical and translational applications. Archives of Plastic Surgery 2013; 40(6):666-75.
- 9. Shin H, Ryu HH, Kwon O, Park BS, Jo SJ. Clinical use of conditioned media of adipose tissue-derived stem cells in female pattern hair loss: a retrospective case series study. Int J Dermatol 2015; 54(6):730-5.
- 10. Hercogova J, Ricceri F, Tripo L, Lotti T, Prignano F. Psoriasis and body mass index. Dermatologic Therapy 2010; 23(2)152-4.

- 11. Alexiades-Armenakas M. A quantitative and comprehensive grading scale for rhytides, laxity, and photoaging. Journal of drugs in dermatology: JDD 2006; 5(8):808-9.
- 12.Isik B, Gurel MS, Erdemir AT, Kesmezacar O. Development of skin aging scale by using dermoscopy. Skin Res Technol 2013; 19(2):69-74.
- 13.Du Plessis JL, Engelbrecht S, Laubscher PJ, Van Aarde MN, Franken A. Dermal exposure and changes in skin barrier function of base metal refinery workers co-exposed to cobalt and nickel. Occupational Health Southern Africa 2013;19(1):8-16.
- 14. Laurent A, Mistretta F, Bottigioli D, Dahel K, Goujon C, Nicolas JF, et al. Echographic measurement of skin thickness in adults by high frequency ultrasound to assess the appropriate microneedle length for intradermal delivery of vaccines. Vaccine 2007; 25(34):6423-30.
- 15.Louis KS, Siegel AC. Cell viability analysis using trypan blue: manual and automated methods. Methods Mol Biol 2011; 740:7-12.
- 16. Chrostowska-Plak D, Reich A, Szepietowski JC. Relationship between itch and psychological status of patients with atopic dermatitis. Journal of the European Academy of Dermatology and Venereology: JAEDV. 2013; 27(2):239-42.